CLINICAL TRIAL: NCT04854967
Title: Post-REcovery LIbEration From Oxygen in Exacerbated COPD (RELIEF)
Brief Title: Pilot Study: Post-Recovery LibEration From Oxygen in Exacerbated COPD
Acronym: RELIEF Pilot
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IIR 17-263
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Lung Diseases; Oxygen Therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either usual care or an oxygen de-implementation intervention. The oxygen de-implementation intervention will consist of: 1) an order to rescind the patient's home oxygen 2) an "unlearning" component targeting provider and patient education and 3) a "substitution" component that introduces alternative evidence-based therapies to treat dyspnea (e.g. teach-to-goal inhaler teaching and pursed lip breathing).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- De-implementation Intervention (Experimental): The oxygen de-implementation intervention will consist of: 1) an order to rescind the patient's home oxygen 2) an "unlearning" component targeting provider and patient education and 3) a "substitution" component that introduces alternative evidence-based therapies to treat dyspnea (e.g. teach-to-goal inhaler teaching and pursed lip breathing).
  Interventions: Other: Rescind home oxygen order; Behavioral: Provider Education; Behavioral: Patient Education; Behavioral: Teach-to-goal inhaler training; Behavioral: Pursed lip breathing
- Usual Care (No Intervention): The patient receives usual care from their assigned clinical provider.

INTERVENTIONS:
Other: Rescind home oxygen order — A note will be entered in the medical record describing the participants randomization into the intervention group. The note will be signed by study staff and will accompany the discontinuation of the patient's home oxygen by a study clinician.
  Other Names: De-implement oxygen order
  Arms: De-implementation Intervention
Behavioral: Provider Education — A note will be entered in the medical record informing the patient's individual medical providers (i.e. primary care provider, pulmonologist) of their randomization into the intervention group. The note will include the evidence-base for oxygen use among patients with COPD.
  Arms: De-implementation Intervention
Behavioral: Patient Education — The patient will receive a patient education page about discontinuation of home oxygen after recovery from a hospitalization that was developed by Consumer Reports in conjunction with the "Choosing Wisely" Campaign.
  Arms: De-implementation Intervention
Behavioral: Teach-to-goal inhaler training — Teach-to-goal (TTG) inhaler training is a patient-centered education strategy that has been shown to decrease inhaler misuse and decrease acute care utilization. The training is tailored to the patient and meets guideline recommendations for assessment and instruction of inhaler technique. The rounds of assessment and demonstration can be completed until acceptable skill level is attained and tailored to the specific medication prescribed.
  Other Names: TTG
  Arms: De-implementation Intervention
Behavioral: Pursed lip breathing — Pursed lip-breathing will be taught to the participants randomized to the intervention arm. This simple technique relieves breathlessness and has been shown to improve functional capacity in patients with COPD. Participants will be given an instructional handout to refer to after the visit.
  Arms: De-implementation Intervention

SUMMARY:
The investigators want to decrease inappropriate oxygen use for patients with COPD. The investigators are testing a new program that will stop oxygen prescriptions for patients that no longer need it and will instead provide them with training in skills that have been shown to help patients breathe better. Participants will be randomly assigned to receive the intervention program or usual care. After 12 weeks the investigators will determine if the program helped stop unnecessary oxygen prescription. The investigators will also determine if health status, distance walked during six minutes, and symptoms of breathlessness after walking are different between participants who received the program and those who did not. The investigators will meet with participating patients and their providers after the study is complete to find out how they feel about this program and if it would be possible to put this change into practice.

DETAILED DESCRIPTION:
The purpose of this pilot study is to test an intervention designed to decrease inappropriate oxygen use for patients with COPD. Participants will be randomized to usual care vs. an oxygen de-implementation intervention. Patients assigned to the oxygen de-implementation intervention group will have their active oxygen prescription discontinued, be educated on pursed lip breathing and receive inhaler training. A follow-up assessment will occur at 12 weeks. The primary outcome at 12 weeks will be discontinuation of oxygen. Secondary outcomes include health status as measured by the Clinical COPD Questionnaire (CCQ), tele-six minute walk test (6MWT) distance, and Borg dyspnea scale assessed after the tele-6MWT. Among the intervention group, the investigators will also assess acceptability and feasibility of the intervention for patient participants and their providers.

Recruitment was expected to begin in November 2021 but was delayed due to the COVID-19 Omicron outbreak. Recruitment officially began on April 18, 2022.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Diagnosis of COPD
* Discharged within the past 3 months after hospitalization for COPD exacerbation, CHF exacerbation and/or Pneumonia and Active prescription for supplemental oxygen within 48 hours of discharge that remains active; or Stable COPD with no chronic resting hypoxemia and an active prescription for supplemental oxygen.
* No inpatient or outpatient exacerbations of COPD within the last 30 days
* Smoked at least 10 pack-years of cigarettes
* Room air resting saturation >88% on room air
* Spirometry consistent with COPD (FEV1/FVC < 0.70) and/or evidence of emphysema on CT scan
* Willingness on the part of the participant to stop oxygen if randomized to the intervention
* Ability and willingness to participate in virtual video visits with study staff using VA approved software
* Informed consent for participation

Exclusion Criteria:

* Desaturation during 6MWT <80% for one minute or more
* Non-COPD lung disease that affects oxygenation or survival (including pulmonary hypertension)
* Prescription of oxygen for alternative condition (e.g. bleed-in with positive airway pressure therapy for obstructive sleep apnea)
* Diagnosis expected to result in death in six months or enrollment in hospice
* Participation in another intervention trial
* Cognitive issues that would preclude participation (dementia, stroke, etc.)
* Residence in skilled nursing facility
* Inability to speak, read, or understand English
* Any safety concerns
* Participants clinical team excludes the participant from recruitment or evaluation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Discontinuation of Oxygen at 12 weeks | 12 weeks
  The investigators will assess the proportion of participants who have no active prescription for oxygen at 12 weeks.

SECONDARY OUTCOMES:
Clinical COPD Questionnaire (CCQ) Total Score | Through study completion, an average of 12 weeks
  The disease-specific health status will be measured by the Clinical COPD Questionnaire (CCQ) total Score. The measurement will be defined as the total score of the CCQ at 12 weeks. The CCQ was developed to assess symptoms, functional status, and COPD control and has been used in clinical trials to assess disease specific health status. The measure has strong internal consistency, reliability and validity, and is responsive to change over short time periods. The CCQ consists of 10 items grouped into three domains (symptoms, functional status and mental state), and one total score. Responses range from 0 (never) to 6 (almost all the time). The total score is calculated by adding all the responses and dividing by the total number of items to produce a final score that ranges from 0-6.
tele-six minute walk test distance (tele-6MWT) | Through study completion, an average of 12 weeks
  The total distance walked during 6 minutes at the 12 week virtual visit. Participants will be asked to walk for 6 minutes following a premeasured course which was used at the in-person visit and then given to them to take home for the virtual visit.
Post tele-six minute walk test (tele-6MWT) Borg Dyspnea scale | Through study completion, an average of 12 weeks
  The Borg dyspnea scale assesses the difficulty that a patient is having with breathing at the current moment, and ranges from 0 (nothing at all) to 10 (maximal). Within one minute of completing the tele-6MWT, the participant will be asked to grade the severity of their dyspnea based on the modified Borg dyspnea scale.
Cost of intervention | At study completion, an average of 12 weeks
  The estimate of costs related to the intervention will be obtained by tracking duration of intervention content and processes. The duration of tasks related to identification and evaluation of subject, enrollment and the intervention will be collected. These tasks will be broken down by level of skill required and a cost estimate calculated.
Proportion of potentially eligible participants randomized | At study completion, an average of 12 weeks
  Proportion of potentially eligible participants that are successfully randomized into the study
Proportion of randomized participants completing 12 week follow up | At study completion, an average of 12 weeks
  We will calculate the proportion of randomized patients who complete the 12-week follow-up
Proportion of participants completing in-home spirometry | At study completion, an average of 12 weeks
  The proportion of participants who are able to successfully complete in-home spirometry with coaching by study staff will be assessed at the end of the study.
Proportion of participants completing tele-6MWT | At study completion, an average of 12 weeks
  The proportion of participants who are able to complete the tele-6MWT will be calculated.
Rate of completion of all visits | Through study completion, an average of 12 weeks
  We will assess the rate of completion of all study visits among randomized participants.
Acceptability to patients | At study completion, an average of 12 weeks
  Among intervention participants, we will perform semi-structured interviews to assess acceptability of the oxygen de-implementation intervention to patients.
Acceptability to providers | At study completion, an average of 12 weeks
  Among providers of intervention participants, we will perform semi-structured interviews to assess acceptability of the oxygen de-implementation intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Cecere Feemster, MD MS, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No